CLINICAL TRIAL: NCT03767244
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study of Apalutamide in Subjects With High-risk, Localized or Locally Advanced Prostate Cancer Who Are Candidates for Radical Prostatectomy
Brief Title: A Study of Apalutamide in Participants With High-Risk, Localized or Locally Advanced Prostate Cancer Who Are Candidates for Radical Prostatectomy
Acronym: PROTEUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108535; 56021927PCR3011 (Other: Janssen Research & Development, LLC); 2018-001746-34 (EudraCT Number); 2023-506153-38-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apalutamide + ADT (Experimental): Participants will receive androgen deprivation therapy (ADT) plus oral administration of apalutamide 240 milligram (mg) (4 tablets of 60 mg each) daily in each cycle (each cycle of 28 days). Participants will receive six cycles of treatment, followed by radical prostatectomy (RP) with pelvic lymph node dissection (pLND), followed by an additional six cycles of treatment. A Long-Term Extension (LTE) may be initiated at sponsor's discretion after completion of the primary endpoint analysis.
  Interventions: Drug: Apalutamide; Drug: Androgen Deprivation Therapy (ADT)
- Placebo + ADT (Experimental): Participants will receive ADT with oral administration of matching placebo treatment daily in each cycle (each cycle of 28 days). Participants will receive six cycles of placebo treatment, followed by RP with pLND, followed by an additional six cycles of placebo treatment. A LTE may be initiated at sponsor's discretion after completion of the primary endpoint analysis.
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Placebo

INTERVENTIONS:
Drug: Apalutamide — Participants will receive apalutamide 240 mg (4 tablets of 60 mg each) orally once daily.
  Other Names: JNJ-56021927
  Arms: Apalutamide + ADT
Drug: Androgen Deprivation Therapy (ADT) — Participants will receive a stable regimen of ADT - gonadotropin-releasing hormone analog (agonist or antagonist) (GnRHa). ADT is a kind of hormone therapy for prostate cancer. GnRHa will be administrated to achieve and maintain sub-castrate concentrations of testosterone (50 nanogram per deciliter [ng/dL]).
Drug: Placebo — Participants will receive matching placebo oral tablets daily.
  Arms: Placebo + ADT

SUMMARY:
The purpose of this study is to determine if treatment with apalutamide plus androgen deprivation therapy (ADT) before and after radical prostatectomy (RP) with pelvic lymph node dissection (pLND) in participants with high-risk localized or locally advanced prostate cancer results in an improvement in pathological complete response (pCR) rate and metastasis-free survival (MFS) as compared to placebo plus ADT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* High-risk disease defined by a total Gleason Sum Score greater than equal to (>=) 4+3 (=Grade Groups [GG] 3-5) and >=1 of the following 4 criteria: a) Any combination of Gleason Score 4+3 (= 3) and Gleason Score 8 (4+4 or 5+3) in >= 6 systematic cores (with >=1 core Gleason Score 8 [4+4 or 5+3] included); b) Any combination of Gleason Score 4+3 (=GG 3) and Gleason Score 8 (4+4 or 5+3) in >=3 systematic cores and Prostate-specific antigen (PSA) >=20 ng/mL (with >= 1 core Gleason Score 8 [4+4 or 5+3] included); c) Gleason Score >=9 (=GG 5) in at least 1 systematic or targeted core; d) At least 2 systematic or targeted cores with continuous Gleason Score >=8 (=GG 4), each with > 80 percent (%) involvement
* Candidate for radical prostatectomy with pelvic lymph node dissection as per the investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Contraceptive use by male participants (and female partners of male participants enrolled in the study who are of childbearing potential or are pregnant) should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies
* Able to receive androgen deprivation therapy (ADT) for at least 13 months

Exclusion Criteria:

* Distant metastasis based on conventional imaging (clinical stage M1). Nodal disease below the iliac bifurcation (clinical stage N1) is not an exclusion. Diagnosis of distant metastasis (clinical M stage; M0 versus M1a, M1b, M1c) and pelvic nodal disease (clinical N stage; N1 versus N0) will be assessed by central radiological review. Participants are considered eligible only if the central radiological review confirms clinical stage M0
* (a) Prior treatment with androgen receptor antagonists; (b) Treatment with gonadotropin-releasing hormone analog (GnRHa) prior to informed consent form (ICF) signature
* History of prior systemic or local therapy for prostate cancer, including pelvic radiation for prostate cancer
* Use of any investigational agent less than or equals to (<=)4 weeks prior to randomization or any therapeutic procedure for prostate cancer at any time
* Major surgery <=4 weeks prior to randomization
* Any of the following within 12 months prior to first dose of study drug: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (example, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias or New York Heart Association Class II to IV heart disease; uncomplicated deep vein thrombosis is not considered exclusionary

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2517 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2028-10-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Pathologic complete response (pCR) | Approximately 4 years
  pCR is assessed by a pathology blinded independent central radiology review (BICR) as defined in the pathology charter.
Metastasis-Free Survival (MFS) | Up to 7 years and 5 months
  MFS is defined as the time from randomization to the date of the occurrence of radiographic distant metastasis evaluated by radiology BICR, incidental pathologic finding of distant metastasis, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Prostate Specific Antigen (PSA)-Free Survival | Approximately 4 years
  PSA-free survival with testosterone recovery defined as the time from randomization to the first detectable serum PSA level with recovered testosterone levels after undetectable PSA post-radical prostatectomy with pelvic lymph node dissection or death, whichever occurs first.
Event Free Survival (EFS) | Up to 7 years and 5 months
  EFS defined as time from randomization to any of the following events: biochemical failure (BCF); or local or regional recurrence by BICR or histopathological assessment; or distant metastasis by BICR or histopathological assessment; or death.
Time to Subsequent First Treatments (TTST-1) | Up to 7 years and 5 months
  TTST-1 is defined as the time from randomization to the date of first subsequent therapy.
Time to Distant Metastasis (TTDM) | Up to 7 years and 5 months
  TTDM is defined as the time from the date of enrollment until the first date of distant metastasis.
MFS Based on Conventional Imaging | Up to 7 years and 5 months
  MFS based on conventional imaging, defined as the time from randomization to the date of the first occurrence of radiographic distant metastasis on CT/MRI and bone scan by radiology BICR, pathologic finding of distant metastasis, or death from any cause, whichever occurs first.
Number of Participants with No Evidence of Disease (NED) at 4 Years | Up to 4 years
  Number of participants with NED at 4 years will be reported. NED at 4 years is defined as: (a) alive, (b) Undetectable prostate-specific antigen (PSA), (c) No distant metastasis, (d) No local or regional recurrence, (e) No subsequent therapy for prostate cancer, (f) Testosterone recovery to physiological testosterone levels, defined as 200 nanograms per deciliter (ng/dL).
Number of Participants with Vital Signs Abnormalities as a Measure of Safety and Tolerability | Up to 30 days after last dose of study drug (Approximately 8 years)
  Number of participants with vital signs (including body temperature, heart rate, respiratory rate, and blood pressure) abnormalities will be reported.
Number of Participants with Physical Examinations Abnormalities as a Measure of Safety and Tolerability | Up to 30 days after last dose of study drug (Approximately 8 years)
  Number of participants with physical examinations (including general appearance of the participant, height, weight, and examination of the skin, ears, nose, throat, lungs, heart, abdomen, extremities, musculoskeletal system, lymphatic system, and nervous system) abnormalities will be reported.
Number of Participants with Laboratory Abnormalities as a Measure of Safety and Tolerability | Up to 30 days after last dose of study drug (Approximately 8 years)
  Blood samples for serum chemistry and hematology will be collected at predefined time points for clinical laboratory testing.
Number of Participants with Treatment Compliance Rate | Up to 30 days after last dose of study drug (Approximately 8 years)
  Number of participants who are complaint with study treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (202):
- United States (44):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine Medical Center Chao Family Comprehensive Cancer Center, Orange, California
  - UC Davis Medical Center, Sacramento, California
  - AdventHealth Medical Group Urology of Denver, Denver, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - Urology Specialists LLC, Hialeah, Florida
  - Mayo Clinic - Division Of Hematology/oncology, Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health / Baptist Health Medical Group, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Ochsner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Michigan Institute of Urology, PC, Troy, Michigan
  - Saint Louis University, St Louis, Missouri
  - Urology Cancer Center, PC, Omaha, Nebraska
  - Albany Medical College, Albany, New York
  - Great Lakes Physician PC d/b/a Western New York Urology Associates, Cheektowaga, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Carolina Urology Partners, PLLC, Huntersville, North Carolina
  - Cleveland VA Medical Center, Cleveland, Ohio
  - Oklahoma City VAMC, Oklahoma City, Oklahoma
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - Greenville Health, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - VA North Texas Health Care System, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, PLCC, Virginia Beach, Virginia
  - CAMC Memorial Hospital, Charleston Area Medical Center Physicians, Charleston, West Virginia
- Argentina (6):
  - Hospital Aleman, Caba
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Uroclinica, Mendoza
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Australia (9):
  - Eastern Health - Box Hill Hospital, Box Hill
  - St Vincent s Hospital Sydney, Darlinghurst
  - Austin Health, Heidelberg
  - Australian Urology Associates Pty Ltd, Malvern
  - Royal Melbourne Hospital, Parkville
  - Northern Cancer Institute, St Leonards
  - Sydney Adventist Hospital, Wahroonga
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Brazil (8):
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - Oncosite - Centro de Pesquisa Clínica em Oncologia Ltda, Ijuí
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Universidade do Estado do Rio de Janeiro - UERJ, Rio de Janeiro
  - Associacao Umane, São Paulo
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Instituto Do Cancer Brasil, Três Lagoas
- Canada (8):
  - Prostate Cancer Centre, Calgary, Alberta
  - Vancouver Prostate Centre, Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - London Health Sciences Center, London, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - CHUM - Centre hospitalier universitaire de Montreal, Montreal, Quebec
  - CHU de Quebec Universite Laval Hopital de l Enfant Jesus, Québec, Quebec
- Czechia (6):
  - Fakultni nemocnice Hradec Kralove, Hradec Králove
  - Krajská nemocnice Liberec, Liberec
  - Uromedical Center s.r.o., Olomouc
  - Fakultni nemocnice Plzen, Urologicka klinika, Pilsen
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Thomayerova nemocnice, Prague
- France (11):
  - CHU d'Angers, Angers
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - Hopital Pellegrin CHU Bordeaux, Bordeaux
  - APHP - Hopital Henri Mondor, Créteil
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - CHU de Nantes hotel Dieu, Nantes
  - Institut Mutualiste Montsouris, Paris
  - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - CHRU Tours Hopital Bretonneau, Tours
- Germany (13):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Städtisches Klinikum Braunschweig gGmbH - Standort Salzdahlumer, Braunschweig
  - Universitaetsklinikum Koelnt, Cologne
  - Praxis Dr. med. Ralf Eckert, Eisleben Lutherstadt
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Prostata zentrum Nordwest, Gronau
  - Martini-Klinik am Universitätsklinikum Hamburg-Eppendorf Urologie, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitatsklinikum Schleswig Holstein Campus Lubeck, Lübeck
  - Klinikum St. Elisabeth Straubing GmbH, Straubing
  - Kliniken Nordoberpfalz, Klinik für Urologie, Weiden/Opf
  - Praxisgemeinschaft f. Onkologie u. Urologie - Germany, Wilhelmshaven
- Israel (6):
  - Asaf Harofe Medical Center, Beer Yaakov
  - Rambam Health Care Campus, Haifa
  - Tel Aviv University Sackler School of Medicine - Meir Medical Center (MMC), Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (17):
  - Policlinico Abano Terme, Abano Terme
  - Generale Regionale F. Miulli, Acquaviva delle Fonti
  - Ospedale di Bassano del Grappa, Bassano del Grappa
  - ASST Spedali Civili Brescia, Brescia
  - ASL2 Lanciano - Vasto - Chieti - Ospedale 'SS Annunziata' di Chieti, Chieti
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - San Raffaele Turro - Istituto di Ricovero e Cura a Carattere Scientifico, Milan
  - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Clinica di Urologia Policlinico di Modena - Universita di Modena e reggio Emilia, Modena
  - Università del Piemonte Orientale - Ospedale Maggiore della Carità di Novara, Novara
  - Universita degli Studi di Torino - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
  - Universita Campus Bio-Medico di Roma, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
  - Ospedale Molinette, AO Città della Salute e della Scienza di, Torino
  - UOC di Urologia AOU Integrata di Verona - Polo Chirurgico Confortini - Ospedale Borgo Trento, Verona
- Japan (23):
  - Akita University Hospital, Akita
  - Chiba University Hospital, Chiba
  - Chiba Cancer Center, Chūōku
  - Hakodate Goryoukaku Hospital, Hakodate
  - Hirosaki University Hospital, Hirosaki
  - Kanazawa University Hospital, Kanazawa
  - Kobe City Medical Center General Hospital, Kobe
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Kurume University Hospital, Kurume
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Kitasato University Hospital, Minamiku
  - University of Miyazaki Hospital, Miyazaki
  - Nagano Municipal Hospital, Nagano
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Sakai
  - Toho University Sakura Medical Center, Sakura
  - Hokkaido University Hospital, Sapporo
  - Iwate Medical University Hospital, Shiwa-gun
  - Nippon Medical School Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Yamaguchi University Hospital, Ube
  - Yokohama City University Medical Center, Yokohama
- Netherlands (4):
  - Antoni van Leeuwenhoek, Amsterdam
  - Catharinaziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis (St. Antonius Hospital), Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
- Poland (6):
  - Samodzielny Publiczny Wielospecjalistyczny Zaklad Opieki Zdrowotnej Mswia W Bydgoszczy, Bydgoszcz
  - Szpital Uniwersytecki NR 1 IM Dr Antoniego Jurasza, Bydgoszcz
  - Szpital Wojewodzki im Mikolaja Kopernika w Koszalinie, Koszalin
  - Pratia MCM Krakow, Krakow
  - City Clinic Sp. z o.o., Warsaw
  - Dolnoslaskie Centrum Onkologii, Oddzial Chirurgii Onkologicznej II - Urologia, Wroclaw
- Russia (7):
  - Altai Regional Oncology Dispensary, Barnaul
  - Chelyabinsk Regional Clinical Center Of Oncology And Nuclear Medicine, Chelyabinsk
  - Moscow City Clinical Hospital # 62, Moscow
  - Hertzen Oncology Research Institute, Moscow
  - Clinical Oncology Dispensary, Omsk
  - Medical-sanitary unit 'Neftyanik', Tyumen
  - Vologda Regional Oncological Dispensary, Vologda
- South Korea (5):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (14):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Puerta Del Mar, Cadiz
  - Hosp. Gral. Univ. de Castellon, Castellon
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Fund. Hosp. de Manacor, Manacor
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Inst. Valenciano de Oncologia, Valencia
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - Chi Mei Medical Center Yong Kang, Tainan
  - National Taiwan University Hospital., Taipei
- United Kingdom (9):
  - Southmead Hospital, Bristol
  - University Hospital of Wales, Cardiff
  - Ninewells Hospital, Dundee
  - The Royal Marsden NHS Trust, London
  - University College London, London
  - Lancashire Teaching Hospitals NHS Foundation Trust Royal Preston Hospital, Preston
  - Royal Marsden Hospital, Sutton
  - Mid Yorkshire NHS Trust, Wakefield
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Ravi P, Kwak L, Xie W, Kelleher K, Acosta AM, McKay RR, Kibel AS, Taplin ME. Neoadjuvant Novel Hormonal Therapy Followed by Prostatectomy versus Up-Front Prostatectomy for High-Risk Prostate Cancer: A Comparative Analysis. J Urol. 2022 Oct;208(4):838-845. doi: 10.1097/JU.0000000000002803. Epub 2022 Sep 9. PMID 36082554